CLINICAL TRIAL: NCT01341171
Title: Platelet Modulation in the Control of Angiogenesis: The Impact of Tamoxifen and Aromatase Inhibitors on Platelet Activation and Angiogenic Proteins
Brief Title: The Impact of Tamoxifen and Aromatase Inhibitors on Platelet Proteins
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Chris Holmes, Associate Professor of Medicine, University of Vermont
Other Study IDs: V0805
Record Dates: First submitted 2010-07-07; First posted 2011-04-25 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: tamoxifen; aromatase inhibitors; breast cancer; platelets
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — serum, plasma, platelet activated samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tamoxifen or aromatase inhibitors

SUMMARY:
Single phlebotomy study involving women receiving tamoxifen or aromatase inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* women routinely taking tamoxifen or aromatase inhibitor therapy as prescribed by their oncologist

Exclusion Criteria:

* Use of heparin, warfarin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women using tamoxifen or aromatase inhibitor therapy for greater than 6 months
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Angiogenic Protein levels | following 6 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Chris E Holmes, MD, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States